CLINICAL TRIAL: NCT05500963
Title: Reducing Fatigue in People With Multiple Sclerosis by Treatment With Transcutaneous Electrical Nerve Stimulation
Brief Title: Reducing Fatigue in People With Multiple Sclerosis by Treatment With TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Roger Enoka, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-0394
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Effective dose (Experimental): • The effective dose of TENS will be set at an intensity to elicit slight contractions in each target muscle, as we have done previously. It will be delivered as 5-Hz bursts (7 pulses at 100 Hz/burst) and applied during the light exercises. The applied current (<20 mA) will differ slightly for each of the four muscle groups and will be determined while the person is standing. The current will be set at the beginning of every treatment session for both groups of participants.
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Sham dose (Sham Comparator): • The current intensity for the sham dose will be set at sensory threshold, which will be less than that used for the effective dose. After beginning each exercise set, the current for the sham dose will decay to 0 mA within 30 s. In a preliminary study that included a sham dose of TENS, we found that only two of the experienced dancers in the sham group detected the gradual decline in TENS current from its initial value slightly above motor threshold when performing prescribed exercises.
  Interventions: Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — Electrical stimulation applied over selected leg muscle will activate sensory receptors that will transmit signals back into the central nervous system.

SUMMARY:
The objective of the randomized, sham-controlled trial will be to evaluate the effectiveness of treatment with transcutaneous electrical nerve stimulation (TENS) at reducing the level of fatigue experienced by people with MS.

DETAILED DESCRIPTION:
We will compare the changes in self-reported levels of fatigue (symptom intensity) and measures of fatigability (work capacity) from before to after a 6-week intervention. Participants (18-65 yrs) will be randomly assigned to one of two groups: one group will receive an effective dose of TENS and the other group (control) will be given a sham dose of TENS. The treatment will be applied during 18 sessions (3x/week for 6 weeks) and delivered through electrodes placed on the skin overlying the dorsiflexor (tibialis anterior) and hip flexor (rectus femoris) muscles of both legs. Participants will be evaluated before (Week 0), during (Week 4), and after (Weeks 7 and 11) the 6-week intervention.

Our long-term goal is to develop strategies that can reduce the impact of fatigue on the daily activities of persons with MS. The objective of the randomized, sham-controlled trial will be to evaluate the effectiveness of treatment with TENS at reducing the level of fatigue experienced by people with MS. Our central hypothesis is that treatment with TENS applied to selected leg muscles in people with MS will produce superior improvements in self-reported and measured levels of fatigue and fatigability compared with a sham dose of TENS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women18-65 yrs
* Able to read, understand, and speak English to ensure safe participation in the project
* Clinical diagnosis of relapsing-remitting MS
* Self-reported difficulty with walking
* On stable doses of Ampyra, provigil, or other symptomatic-treating medications
* No relapse or systemic steroids within the last 30 days
* Able to arrange transportation to the Boulder campus

Exclusion Criteria:

* Vision or hearing problems that have not been corrected
* Problems with sensations to temperature, pressure, or pain
* Any arm or leg problems that would influence the ability to hold a weight
* Surgery to the arms or legs that continues to bother the participant
* Metal implants
* Medical diagnosis or condition that is considered to be an absolute or relative contraindication to participating in exercise training, such as major renal, pulmonary, hepatic, cardiac, gastrointestinal, HIV, cancer (other than treated basal cell cancer), other neurological disorders, or pregnancy
* History of head injury or stroke
* Taking antidepressants, anticholinergics, stimulants, sedatives, cannabis, illicit drugs or medications to treat herpes or neurologic pain.
* Diagnosis of diabetes mellitus
* Poorly controlled hypertension
* History of seizure disorders
* ≥2 alcoholic drinks/day, or present history (last 6 months) of drug abuse
* Spasticity that requires the individual to change intended activities more often than once a week
* Skin diseases or sensation problems in the legs or hands that influences some activities more often than once a week
* Inability to attend exercise sessions 3 days per week for 6 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Changes at Weeks 4, 7, and 11
  Questionnaire scores - PROMIS Fatigue (MS) 8a
Walking limitations | Changes at Weeks 4, 7, and 11
  Questionnaire scores - MS Walking Scale-12
Walking endurance | Changes at Weeks 4, 7, and 11
  6-min walk test in meters
Mobility | Changes at Weeks 4, 7, and 11
  Assessment of static and dynamic balance with Mobility Lab, APDM Inc

SECONDARY OUTCOMES:
Quality of life questionnaire | Changes at Weeks 4, 7, and 11
  Questionnaire scores
Muscle strength | Changes at Weeks 4, 7, and 11
  Maximal force in newtons applied by the dorsiflexors and hip flexors of each leg

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Enoka RM, Almuklass AM, Alenazy M, Alvarez E, Duchateau J. Distinguishing between Fatigue and Fatigability in Multiple Sclerosis. Neurorehabil Neural Repair. 2021 Nov;35(11):960-973. doi: 10.1177/15459683211046257. Epub 2021 Sep 28. PMID 34583577
- [Result] Almuklass AM, Davis L, Hamilton LD, Hebert JR, Alvarez E, Enoka RM. Pulse Width Does Not Influence the Gains Achieved With Neuromuscular Electrical Stimulation in People With Multiple Sclerosis: Double-Blind, Randomized Trial. Neurorehabil Neural Repair. 2018 Jan;32(1):84-93. doi: 10.1177/1545968317753681. Epub 2018 Jan 24. PMID 29366377
- [Result] Almuklass AM, Capobianco RA, Feeney DF, Alvarez E, Enoka RM. Sensory nerve stimulation causes an immediate improvement in motor function of persons with multiple sclerosis: A pilot study. Mult Scler Relat Disord. 2020 Feb;38:101508. doi: 10.1016/j.msard.2019.101508. Epub 2019 Nov 6. PMID 31715503
- [Result] Alenazy M, Daneshgar Asl S, Petrigna L, Feka K, Alvarez E, Almuklass AM, Enoka RM. Treatment with electrical stimulation of sensory nerves improves motor function and disability status in persons with multiple sclerosis: A pilot study. J Electromyogr Kinesiol. 2021 Dec;61:102607. doi: 10.1016/j.jelekin.2021.102607. Epub 2021 Oct 13. PMID 34710779